CLINICAL TRIAL: NCT01383902
Title: The Effect of Meal Type on the Rate of Gastric Emptying
Brief Title: Chocolate Meal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Alan Mackie / Research Leader, Institute of Food Research
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: IFR03/2008
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Impact of Food Composition on Gastric Emptying

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dessert / chocolate (Other)
  Interventions: Other: Food type

INTERVENTIONS:
Other: Food type — 1ml, 1ml, 5ml, 50ml, 6ml, 20ml, 60ml and 200ml of chocolate dessert or 1 g, 1 segment (5 segments to a bar) repeated 6 times, 2 bars repeated twice of chocolate bars

SUMMARY:
This comparative pilot study is designed to compare the rates of gastric emptying and by inference rates of digestion of challenge meals. Two types of meal will be compared, chocolate mousse style dessert and chocolate bars. The information from this study will then be compared to the elicitation times for both objective and subjective symptoms in the allergic patients who have been challenged in a different study using the same two meals.

ELIGIBILITY:
Inclusion Criteria:

* Male (hormonal status of women would introduce more variation within small group)
* Age 20-50y
* BMI 19-30
* Nominally healthy
* Normally eat lunch
* Willing to eat dark chocolate bars and chocolate dessert.
* Provides informed written consent

Exclusion Criteria:

* Smokers or smoked within the last year (smoking affects satiety/hunger and volunteer's will not be able to smoke during the study day at the hospital)
* Diagnosed with any long term illness requiring active treatment e.g. diabetes, cancer, cardiovascular disease
* Have had surgery on the stomach or intestine or suffered from gastrointestinal disease.
* Regular (more than once in 10 days) use of antacids, laxatives
* Diagnosis with any mouth, dental, throat or digestive problem that may affect normal eating and digestion of food.
* Volunteers taking part in another study (other than a questionnaire based study).
* Blood pressure greater than 160/100 or less than 90/50 or 95/55 if symptomatic.
* Individuals with special dietary requirements (eg vegetarians)
* People with eating disorders (eg. anorexia, bulimia)
* If any of the clinical screening results are indicative of a health problem which would affect the volunteers well-being or which would affect the study data.
* Refusal to give permission to inform GP of participation in study
* Allergic to any of the constituents of the test meal
* Recent unexplained weight gain or loss
* History of back problems or any other condition which limit ability to repeatedly sit up and lie down
* Hiatus Hernia
* MRI scanning specific exclusion criteria

  * Cardiac pacemaker or artificial heart valve
  * Head surgery or any surgery in the last 6 months
  * Aneurysm clips (metal clips from surgery)
  * Implant, pump or any medical device in the body (eg cochlear implant, neurostimulator, intra-venticular shunt)
  * Worked with metals (using lathes or grinders) or sustained injury to eyes involving metal splinters or fillings
  * Have artificial eyes or limbs
  * Have been injured with shrapnel or bullets
  * Suffer from fits, blackouts or epilepsy
  * Claustrophobia sufferer

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
A series of MRI images of the abdomen giving gastric emptying and layering data | 4 hours
  To produce gastric emptying and layering data from MRI images on healthy volunteers using a nine differing dose protocol in two different foods.

SECONDARY OUTCOMES:
Use of MRI for measuring gastric emptying rates | 4 hours
  An additional underpinning objective is to evaluate and optimise the MRI method for imaging gastric function as a reliable tool for future clinical and nutritional research.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Institute of Food Research, Norwich, Norfolk
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk